CLINICAL TRIAL: NCT01690962
Title: A Nutritional Intervention for Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PCRM DN-1
Record Dates: First submitted 2012-09-17; First posted 2012-09-24 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Diabetic Neuropathy
Keywords: diabetic neuropathy, diet, vegan, vegetarian
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Diet, Vegan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vegan diet and vitamin B12 supplement (Experimental): The diet/supplement group will be asked to follow a low-fat, vegan diet for 20 weeks, and take a vitamin B12 supplement daily.
  Interventions: Other: Vegan diet and vitamin B12 supplement
- Vitamin B12 supplement (Active Comparator): The supplement group will be asked to take a daily vitamin B12 supplement, and to make no changes to their current diet.
  Interventions: Dietary Supplement: Vitamin B12 supplement

INTERVENTIONS:
Other: Vegan diet and vitamin B12 supplement — A low-fat, vegan diet (no meat, fish, eggs or dairy products) and a vitamin B12 supplement in the form of 2000mcg of methylcobalamin
  Other Names: Vegan diet
  Arms: Vegan diet and vitamin B12 supplement
Dietary Supplement: Vitamin B12 supplement — A daily vitamin B12 supplement in the form of 2000mcg of methylcobalamin
  Arms: Vitamin B12 supplement

SUMMARY:
The purpose of this study is to assess whether, in individuals with diabetic neuropathy, a low-fat, vegan diet in combination with a vitamin B12 supplement improves pain, sensation and other subjective symptoms, more effectively than a vitamin B12 supplement with no diet changes. The principal measure is pain as measured by the following assessment tools: Michigan Neuropathy Screening Instrument, Norfolk Quality of Life Questionnaire, Neuropathy Impairment Score - Lower Limbs, Neuropathy Total Symptom Score, Neuropathy Pain Scale, McGill Pain Questionnaire and Global Impression Scale. The study duration is 20 weeks.

This study also examines the effects of a low-fat, vegan diet on mood, using the Center for Epidemiologic Studies Depression Scale-Revised, and the Beck Depression Inventory.

DETAILED DESCRIPTION:
The following determinations will be made at baseline, mid-point, and end of each 20-week study period, as well as at one-year follow up:

General status, symptoms, and medication accounting. Participants will be asked to report changes in their health and medication use.

Disease Activity. The following assessments will be used to measure pain and changes in sensory perception related to diabetic neuropathy:

* Michigan Neuropathy Screening Instrument. The MNSI questionnaire consists of 15 questions followed by a single 8-point clinical examination involving inspection of the foot, assessment of ankle reflexes, and semi-quantitative determination of vibration perception.
* Norfolk Quality of Life Questionnaire Norfolk QOL-DN is a 47-item questionnaire developed by the Eastern Virginia Medical School, Norfolk, VA, for assessing subjects' perception of the effects of diabetes and diabetic neuropathy. It consists of 28 items pertaining specifically to to small fiber, large fiber and autonomic nerve function symptoms, and activities of daily living (ADL).
* Neuropathy Impairment Score for Lower Limbs (NIS-LL) The NIS-LL is the lower limb component of the full Neuropathy Impairment Score (NIS) and has 3 domains including: muscle weakness, reflexes, and sensation. The maximum score is 88 points. Based on experience with and data collected from these clinical trials, the Peripheral Nerve Society considers a 2 point change on the NIS-LL to correspond to a meaningful change in clinical status.
* Neuropathy Total Symptoms Score (NTSS-6) Neuropathy total symptom score-6 (NTSS-6) is a neuropathy sensory symptom scale that is designed to evaluate the frequency and intensity of individual neuropathy sensory symptoms identified frequently by patients with DPN. A total of six questions are synthesized to identify and quantify the specific positive and negative symptoms associated with sensory deficits in patients.
* Neuropathy Pain Scale In order to assess and differentiate qualities of pain, Galer and Jensen developed the Neuropathic Pain Scale (NPS) in 1997. The NPS is composed of 10 items that assess two global pain domains including pain intensity and unpleasantness, and six pain qualities, including sharp, hot, dull, cold, sensitive, and itchy pain, in two dimensions (internal and cutaneous).
* McGill Pain Questionnaire The McGill Pain Questionnaire (MPQ) is used to specify subjective pain experience using sensory, affective and evaluative word descriptors. The short form of the McGill Pain Questionnaire (SF-MPQ) contains 11 questions referring to the sensory dimension of the pain experience and four related to the affective dimension.
* Global Impression Scale Global impression scale (GIS) is also termed global rating of change scales (GRC) and was developed to assess patients' overall improvement or deterioration in a clinical setting, and has been frequently used in musculoskeletal and chronic pain trials.

Height. Height will be measured at baseline (only) with participants standing barefoot with their backs to a wall-mounted stadiometer and heels against the wall, recorded to the nearest 0.5 cm.

Body weight. With participants wearing light, indoor clothing but without shoes, body weight will be measured to the nearest 0.1 kg, using a digital scale.

Blood pressure. A digital blood pressure monitor and a cuff of a size appropriate to the participant's arm will be used. The cuff size for each participant will be recorded for consistency of use at each visit. Participants will be asked to remove all clothing that covers the location of cuff placement and then rest in a seated position for 5 minutes with legs uncrossed, without talking or reading. The back and arm will be supported such that the middle of the cuff on the upper arm is at the level of the right atrium (the mid-point of the sternum). Three measurements will be taken at 1-minute intervals. The first measurement will be disregarded, and the mean of the remaining 2 measurements will be calculated.

Serum cholesterol and triacylglycerol concentrations will be measured using the Olympus Cholesterol Reagent on Olympus Chemistry Analyzers. HDL-cholesterol will be measured directly using the HDL-C plus 3rd generation test with the Roche direct HDL-cholesterol assay.Low density lipoprotein cholesterol (LDL-C) concentration will be estimated using the Friedewald equation. Plasma triglyceride levels will be measured using Olympus Chemistry analyzers from Quest Diagnostics.

Comprehensive Metabolic Panel. These values will be evaluated at baseline, 20 weeks, and one-year follow-up.

Hemoglobin A1c. Hemoglobin A1c will be measured in whole blood using the COBAS INTEGRA on Roche clinical chemistry analyzers.

Glucose. Plasma glucose will be measured using an Olympus Chemistry Analyzer from Quest Diagnostics, Baltimore, MD, USA.

Urinary albumin and creatinine will be assessed on spot urine samples. Samples for the albumin assay will be tested using the K-Assay High-Sensitive Microalbumin assay from Quest Diagnostics.

Apolipoprotein E (APOE): Participants who consent to this aspect of the study will be genotyped for the ε2, ε3, and ε4 alleles. A sample of approximately 5 ml of the participant's blood is required and will be drawn simultaneously with the 20-week health assessment labs. Individuals with diabetes are at greatly increased risk of developing Alzheimer's disease, and some studies have suggested that the effect of saturated fat intake on Alzheimer's risk may be most evident in (or even limited to) carriers of the APOEε4 allele. The ApoE protein produced by the APOE gene is a major plasma apolipoprotein and the primary cholesterol carrier in the brain [62]. As a group, these individuals have higher plasma LDL concentrations, compared with APOEε3 homozygotes [63] Moreover, APOE status may influence the relationship between dietary intake and plasma lipid concentrations [63]. APOE determination may provide useful information as to who benefits from dietary changes that aim to modify plasma lipid concentrations, with implications for subsequent risk of cardiovascular disease and Alzheimer's disease. The blood test will be drawn once, at the 20-week health assessment only. This test will be optional. If participants decide not to do the test, it will not affect their status in the study. The blood samples that are collected will be used for APOE allele testing for this study only. All samples will be destroyed after analysis and no part of the specimen will be retained per policy of Quest Diagnostics.

Genotyping for Taq1 A and Taq1B polymorphisms. Participants who consent to this aspect of the study will be genotyped for the A1 and B1 alleles, using the PCR method [64] A sample of approximately 5 ml of the participant's blood is required and will be drawn simultaneously with the 20-week health assessment labs. Studies suggest that the A1 allele of the Taq1A polymorphism (rs1800497), located ≈10 kb downstream of the D2 dopamine receptor (DRD2) gene, may influence dietary behavior and response to treatment. Individuals with the A1 allele generally have a lower-than-normal complement of dopamine receptors (DRD2) in the human brain, and are more likely than others to engage in smoking, substance abuse, and compulsive gambling [65]. The prevalence of A1 and B1 alleles of the DRD2 gene is strongly associated with severe alcoholism [66]. Further, the A1 allele is also common among obese individuals [67]. We identified this allele in approximately half of individuals with type 2 diabetes participating in a research study [68]. The possibility that genetic factors may influence dietary behavior may mean that extended support is essential for facilitating dietary transitions among many, if not all, individuals with diabetes. In group settings, support can be engaging and cost effective. The blood test will be drawn once, at the 20-week health assessment only. This test will be optional. If participants decide not to do the test, it will not affect their status in the study. The blood samples that are collected will be used for TaqA1 allele testing for this study only. All samples will be destroyed after analysis and no part of the specimen will be retained per policy of The Biological Samples Processing Core Facility (BSPC) at the University of California, Los Angeles (UCLA).

Skin biopsy. A single skin biopsy (3 millimeters in diameter and 4 millimeters in depth) will be removed from one of three sites on the leg at baseline and 20 week health assessment, as well as at one year follow up. The epidermal nerve fiber density test is the only objective test currently available for assessing small fiber neuropathy. A physician or experienced health care professional will clean the skin with alcohol pads and anaesthetize the skin by administering 2% lidocaine with epinephrine. The biopsy will be performed using a 3mm disposable, circular punch. The biopsies will be immediately placed in a fixative container, and then placed into a cooler with an ice pack. The samples will then be shipped for analysis.

2-day dietary record: A 2-day dietary record will be used to assess macro- and micronutrient intakes. Participants will be given the option to complete a manual or online version (online: http://riskfactor.cancer.gov/tools/instruments/asa24/) for collecting and calculating diet and nutrient intake. Participants will need Internet access if they choose to do an online version. If necessary, digitized records will be analyzed using Nutrition Data Systems for Research software (University of Minnesota), by a registered dietitian certified by the Nutrition Coordinating Center.

24-Hour Multi-Pass Dietary Recalls. At weeks 3 and 12, a registered dietitian will make unannounced telephone calls to each participant to administer a 24-hour diet recall, using a multi-pass approach (Nutrition Coordinating Center, University of Minnesota, Minneapolis, MN). These recalls will not be subjected to statistical analysis, but will allow the investigators to check for poor adherence. The ASA-24 is a software tool developed by National Cancer Institute. It enables automated and self-administered 24-hour dietary recalls. The format and design of ASA-24 are based on a modified version of the interviewer-administered Automated Multiple Pass Method (AMPM) 24-hour recall developed by the U.S. Department of Agriculture. Participants will be provided a user name, password, and link to the ASA-24 online diet recall Web site.

The Eating Inventory is a highly reliable 51-item questionnaire providing quantitative measures of dietary restraint, disinhibition, and hunger. It will serve as a gauge of ease in adapting to the intervention diet.

The International Physical Activity Questionnaire short form assesses recent physical activity patterns. The method is highly reliable; an assessment of test-retest repeatability produced a correlation of 0.8.

The Clinical Epidemiologic Studies Depression Scale-Revised (CESD-R) assesses mood. The CES-D is a 20-item self-report measure designed originally for use among the general population. It measures the frequency with which participants have experienced a specific symptom within the preceding week, using a four-point rating scale.

The Beck Depression Inventory II (BDI-II) assesses mood. It is the most widely used instrument for detecting depression. The questions on the BDI-II are in alignment with DSM-IV criteria. Each item is a list of four statements arranged in increasing severity about a particular symptom of depression.

Overall quality of life will be assessed using the SF-36, which is a brief health survey with 36 questions. The SF-36 provides psychometrically-based physical and mental health summary measures. The SF-36 is a general measure that has been administered across various age groups, disease spectra, and treatment regimens. Items on the SF-36 are scored on a scale of 0-100, with a higher score indicating better health-related quality of life.

Medications. Participants in both groups will be asked to keep their medications constant and to add no new nutritional supplements to their current medication regimen, except as recommended by their personal physicians.

The interventions for the diet and supplement group and supplement-only group are described below:

* The diet and supplement group will be asked to follow a low-fat, vegan diet and take a daily vitamin B12 supplement of 1000mcg of methylcobalamin for 20 weeks. According to the American Dietetic Association, vegan and vegetarian diets meet all nutritional requirements when appropriately planned.The diet consists of whole grains, vegetables, legumes, and fruits, with no restriction on energy intake. Animal products, added oils, and sugars will be excluded. In choosing grain products and starchy vegetables (e.g., bread, potatoes), participants will be encouraged to select those retaining their natural fiber and having a glycemic index <70, using tables standardized to a value of 100 for glucose. No meals will be provided. Participants will handle their own food preparation and purchases, with guidance from the research team.
* Participants will be provided with a commercially available supplement containing vitamin B12 and asked to take it daily during the study. Should they wish to continue the diet thereafter, they will be counseled to use any standard multivitamin or other reliable source of vitamin B12.
* The supplement-only group will follow an unrestricted diet, but will be given the identical vitamin B12 supplement of 1000mcg of methylcobalamin as the diet group.

Before randomization, participants will be told that they will either be assigned to a diet and supplement intervention group or a supplement-only group.

For both groups, alcoholic beverages will be limited to one per day for women, and two for men.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 - 65 years old
* A diagnosis of type 2 diabetes
* A diagnosis of diabetic neuropathy for at least 6 months or symptoms of diabetic neuropathy for at least 6 months
* Score of greater than 2 on the Michigan Neuropathy Screening Instrument
* Score of greater than 6on the Norfolk Quality of Life Questionnaire
* Score of greater than 2 on the Neuropathy Impairment Score for Lower Limbs (NIS-LL)
* Score of greater than 1 on the Neuropathy Total Symptom Score 6 (NTSS-6)

Exclusion Criteria:

* Vitamin B12 deficiency
* Alcohol consumption of more than 2 drinks per day or the equivalent, episodic increased drinking (e.g., more than 2 drinks per day on weekends), or a history of alcohol abuse or dependency followed by any current use
* Use of recreational drugs in the past 6 months (past drug use, if fully recovered, is not a criteria for exclusion)
* Pregnancy
* Unstable medical or psychiatric illness
* Likely to be disruptive in group sessions (as determined by research staff)
* Already following a low-fat, vegan diet
* Lack of English fluency
* Inability to maintain current medication regimen
* Inability or unwillingness to participate in all components of the study
* Sensitivity to lidocaine or epinephrine (or their preservatives)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Pain | 20 weeks
  Pain will be measured follow the baseline and 20 week score using n the following assessment tools:
  * Michigan Neuropathy Screening Instrument
  * Norfolk Quality of Life Questionnaire
  * Neuropathy Impairment Score - Lower Limbs
  * Neuropathy Total Symptom Score 6
  * Neuropathy Pain Scale
  * McGill Pain Questionnaire
  * Global Impression Scale
Sensation | 20 weeks
  Sensation will be measured follow the baseline and 20 week score using the following assessment tools:
  * Michigan Neuropathy Screening Instrument
  * Norfolk Quality of Life Questionnaire
  * Neuropathy Impairment Score - Lower Limbs
  * Neuropathy Total Symptom Score 6
Disease activity | 20 weeks
  Disease activity will be measured by change in small fiber density of lower limbs as measured by skin biospy done at baseline and 20 weeks.
Glycemic control | 20 weeks
  Glycemic control will be measured by change in hemoglobin A1c percentage points at baseline and 20 weeks.
Mood | 20 weeks
  Mood will be measured by change in score using the following assessment tools at baseline and 20 weeks:
  * Beck Depression Inventory
  * Center for Epidemiologic Studies Depression Scale Revised

SECONDARY OUTCOMES:
Quality of life | 20 weeks
  Quality of Life will be measured by change in score using the following assessment tools at baseline and 20 weeks:
  * Norfolk Quality of Life Questionnaire
  * MOS SF-36 Questionnaire

OTHER OUTCOMES:
Acceptability of vegan diet | 20 weeks
  Acceptability of vegan diet will be measured by change in score at baseline and 20 weeks using the Eating Inventory questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Barnard, MD, Principal Investigator — Physicians Committee for Responsible Medicine
Locations (1):
- Physicians Committee for Responsible Medicine, Washington D.C., District of Columbia, United States